CLINICAL TRIAL: NCT02839980
Title: Comparative Microbial Epidemiology and Chlorhexidine Suscebtibily of Oropharyngeal and Intestinal Colonization of Hospital Subjects
Brief Title: Microbial Epidemiology and Chlorhexidine Suscebtibily of Oropharyngeal and Intestinal Colonization
Acronym: OroColi
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI15006
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Oropharyngeal Gram-negative Bacilli Colonization
Keywords: oropharyngeal colonization

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- orthopedics (gr1) surgery: parient admitted to the orthopedics (gr1) surgery ward for an elective or semi-emergent surgical procedure.
- thoracic (gr2) surgery: parient admitted to the thoracic (gr2) surgery ward for an elective or semi-emergent surgical procedure.
- abdominal (gr3) surgery: parient admitted to the abdominal (gr3) surgery ward for an elective or semi-emergent surgical procedure.
- ICU (gr4): patients admitted to the ICU with an antcipated length of stay of 3 days or more

SUMMARY:
In this prospective observational multicenter study we aim to determine the prevalence of oropharyngeal and rectal Gram-negative bacilli colonization in 4 population of hospitalized subjects, and their susceptibility to chlorehexidine. We plan to recruit 300 subjects in surgical wards (100 in orthopedics, 100 in thoracic and vascular, 100 in abdominal surgery) and 100 in the ICU. Secondary endpoints are to determine the incidence of the acquisition of such colonization in a 10-day timeframe; determine the phylogentic characteristics of E. coli isolates; to compare the phylogentic characteristics of oropharyngeal and rectal E. coli isolates; to compare the phylogentic characteristics of colonization and potential E. coli infection isolates; to compare the rectal and oropharyngeal colonization composition; description of oropharyngeal microbiote

DETAILED DESCRIPTION:
In this prospective multicenter observational study we aim to determine the prevalence of oropharyngeal and rectal Gram-negative bacilli colonization in 4 population of hospitalized subjects, and their susceptibility to chlorehexidine. We plan to recruit 300 subjects in surgical wards (100 in orthopedics, 100 in thoracic and vascular, 100 in abdominal surgery) and 100 in the ICU. Each participant will undego a oropharyngeal swab collection at day 0, day 5 and day 10 (or discharge), and a rectal swab at day 0 and day 10 or hospital discharge. The Gram-negative bacilli colonization will be identified, E. coli isolates will be studied in terms of phylogeny, antimicrobial and chlorhexidine susceptibility. The primary endpoint is to determine the prevalence of oropharyngeal and rectal Gram-negative bacilli colonization. The secondary endpoints are to determine the incidence of the acquisition of such colonization in a 10 days timeframe; to determine the phylogentic characteristics of E. coli isolates; to compare the phylogentic characteristics of oropharyngeal and rectal E. coli isolates; to compare the phylogentic characteristics of colonization and potential E. coli infection isolates; to compare the rectal and oropharyngeal colonization composition; description of oropharyngeal microbiote.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* admitted in one of the participating surgery wards for elective or semi-emergent surgerical procedure or in one of the ICUs;
* for an anticipated length of stay of 72h

Exclusion Criteria:

* personal history of neck or face irradiation
* bronchectasis;
* patient's or proxies' opposition to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in wards in which emergence of multi-drug resistant bacteria justifies a regular monitoring (i.e. surgical wards and ICU)
Sampling Method: Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2016-10-06 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
proportion of patients with a gram-negative colonization at admission | day 1
  proportion of patients in whom admission oropahryngeal sample will contain at least one gram-negative bacilli among Haemophilus influenzae, an enterobacteria, or a non-fermenting GNB.

SECONDARY OUTCOMES:
incidence of the acquisition of a oropharyngela or rectal GNB colonization | during hospital stay or 10 days if still hospitalized
  incidence of the acquisition of a oropharyngela or rectal GNB colonization in the 4 populations
comparison of the predominant fecal flora with GNB oropharyngeal colonization | hospital stay or 10 days if still hospitalized
characterization of antimicrobial and chlorhexidine susceptibility of gram-negative isolates from oropharyngeal colonization | hospital stay or 10 days if still hospitalized
phylogenetic and virulence factor content of E. coli oropharyngeal and rectal colonization | hospital stay or 10 days if still hospitalized
comparision of the genetic identity of the dominant E. coli rectal and orpohayrngeal colonization with potential nosocomial infections | hospital stay or 10 days if still hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan MESSIKA, MD,, Principal Investigator — Hopital Louis Mourier - Assistance Publique Hopitaux de Paris
Locations (1):
- AP-HP, Louis Mourier Hospital, Colombes, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided